CLINICAL TRIAL: NCT03716505
Title: A Randomized, Multicenter, Double-blind, Parallel, Sham-controlled Study of Non-invasive Vagus Nerve Stimulation for the Prevention of Migraines. (Premium II)
Brief Title: Non-invasive Vagus Nerve Stimulation for the Prevention of Migraines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GM-US-10
Record Dates: First submitted 2018-10-10; First posted 2018-10-23 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Migraine Disorders
Keywords: Prevention; Episodic; Chronic
MeSH Terms: conditions — Migraine Disorders; Recurrence; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Two parallel groups, gammaCore®-Sapphire (active treatment) and a sham (inactive) treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two parallel groups, gammaCore®-Sapphire (active treatment) and a gammaCore®-Sapphire sham (inactive) treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- gammaCore Sapphire active (Active Comparator): Treatment 3 times per day, every day for the 12-week treatment period
  Each of the 3 daily treatments comprises 2 consecutive 120-second stimulations on 1 side, ipsilateral (2 stimulations) to the side of predominate pain, upon waking, lunch time (i.e., between 11:00 AM and 2:00 PM), and prior to sleep, for a total of 6 stimulations per day
  Interventions: Device: gammaCore Sapphire active
- gammaCore Sapphire Sham (Sham Comparator): Treatment 3 times per day, every day for the 12-week treatment period
  Each of the 3 daily treatments comprises 2 consecutive 120-second stimulations on 1 side, ipsilateral (2 stimulations) to the side of predominate pain, upon waking, lunch time (i.e., between 11:00 AM and 2:00 PM), and prior to sleep, for a total of 6 stimulations per day
  Interventions: Device: gammaCore Sapphire Sham

INTERVENTIONS:
Device: gammaCore Sapphire active — GammaCore Sapphire™ is a handheld, non-invasive, low voltage electrical device which stimulates the vagus nerve by producing weak 120 second electrical stimulation cycles that may help reduce, ease, lessen or stop your migraine symptoms. GammaCore Sapphire™ has been approved for the treatment of headache, including migraine by the United States Food and Drug Administration (FDA).
  Arms: gammaCore Sapphire active
Device: gammaCore Sapphire Sham — The sham device is a hand-held portable device that appears identical to gammaCore Sapphire, in look, weight, visual and audible feedback, user application, and control. Like gammaCore Sapphire, the sham device is a multi-use device.
  Arms: gammaCore Sapphire Sham

SUMMARY:
The purpose of the study is to investigate if the use of gammaCore Sapphire™ device reduces the number of migraines preventatively.

DETAILED DESCRIPTION:
The study is a prospective randomized, multi-center, double-blind, parallel, sham-controlled study, designed for comparison of two parallel groups, gammaCore®-Sapphire (active treatment) and a sham (inactive) treatment.

The study period will begin with a four-week run-in period, during which there is no investigational treatment. The purpose of the run-in period will be to establish a baseline of the subject's headache/migraine history for longitudinal comparison.

The run-in period will be followed by a 12-week randomized period when the subjects will be randomized (1:1) to either active treatment or sham (inactive) treatment.

Subjects will dose themselves 3 times per day for 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Between the ages of 18 and 75 years
* Been previously diagnosed with migraine (with or without aura), in accordance with the ICHD-3 criteria
* Experiences between 8 to 20 headaches days per month (during the last 3 months), with at least 5 of them being migraine days
* Onset of migraine at age 50 years or younger
* Agrees to refrain from initiating or changing any prophylactic medications for indications other than migraine

Key Exclusion Criteria:

* Concomitant medical condition that will require oral or injectable steroids during the study
* Currently on a stable regime of more than 1 migraine preventative therapy
* Other significant pain problem (e.g., cancer pain, fibromyalgia, other head or facial pain disorder)
* Known or suspected severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure)
* Known or suspected cerebrovascular disease
* Previous cervical vagotomy
* Currently implanted with an electrical and/or neurostimulator device
* Been implanted with metal cervical spine hardware or has a metallic implant near the nVNS stimulation site
* Known history or suspicion of secondary headache
* Currently using marijuana (including medical marijuana) or has used marijuana (including medical marijuana) or cannabidiol oil within the last 6 months
* Currently takes simple analgesics or NSAIDs >15 days per month or triptans, ergots, or combined analgesics >10 days per month for headaches or other body pain
* Currently takes prescription opioids more than 2 days per month for headaches or body pain
* Failed an adequate trial (2 months or greater) of at least 3 classes of a drug therapy for migraine prevention
* Surgery for migraine prevention
* Undergone nerve block (occipital or other) in the head or neck within the last 3 months
* Received Botox or CGRP mAb injections within the last 6 months
* Pregnant or thinking of becoming pregnant during the study period, or of childbearing years and unwilling to use an accepted form of birth control
* Previously used gammaCore

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Safety and effectiveness of gammaCore Sapphire as a treatment for the prevention of a migraine during the double-blind period measured by Incidence of Unexpected Adverse Events. | 12 weeks
  The primary outcome measurement for effectiveness is the difference between the active and sham treatment groups in the mean reduction in number of migraine days during the last 4 weeks of the 12-week double-blind period (versus during the 4-week run-in period).

SECONDARY OUTCOMES:
Responder rate in the nVNS group compared to the sham group | Last 4 weeks of the 12 week double-blind
  A subject who reports at least a 50% decrease in the number of migraine days during the last 4 weeks in the 12-week double-blind period
Mean reduction in the number of headache days | Last 4 weeks of the 12 week double-blind
  Difference between the nVNS and sham treatment groups in mean reduction in the number of headache days during the last 4 weeks of the 12-week double-blind period
Mean reduction in days on which acute migraine medication | Last 4 weeks of the 12 week double-blind
  Difference between the nVNS and sham treatment groups in the mean reduction in days on which acute migraine medication was taken during the last 4 weeks of the 12 week double-blind period

CONTACTS AND LOCATIONS:
Overall Officials: Peter Staats, MD, Study Director — Chief Medical Officer
Locations (30):
- United States (30):
  - Mayo Clinic, Scottsdale, Arizona
  - The Research Center of Southern California, Carlsbad, California
  - Stanford University Medical Center Hoover Pavilion, Palo Alto, California
  - UCSF Headache Center, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Summit Headache and Neurologic Institute, PC, Englewood, Colorado
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Hartford HealthCare Headache Center, West Hartford, Connecticut
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - NorthShore Ambulatory Care Center, Glenview, Illinois
  - Norton Neurology, Louisville, Kentucky
  - Crescent City Headache and Neurology Center, Chalmette, Louisiana
  - Ochsner North Shore Medical Center, Covington, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan Head Pain & Neurological Institute (MHNI), Ann Arbor, Michigan
  - Headache Neurology Research Institute, Ridgeland, Mississippi
  - StudyMetrix, LLC, City of Saint Peters, Missouri
  - Clinvest Research, Springfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dent Neurologic Institute, Amherst, New York
  - NY Neurology Associates, New York, New York
  - Island Neurological Associates, Plainview, New York
  - Montefiore Headache Center, The Bronx, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - ClinPoint Trials LLC, Waxahachie, Texas
  - Medstar Georgetown University Hospital, McLean, Virginia
  - West Virginia University Hospitals - Department of Neurology, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Najib U, Smith T, Hindiyeh N, Saper J, Nye B, Ashina S, McClure CK, Marmura MJ, Chase S, Liebler E, Lipton RB. Non-invasive vagus nerve stimulation for prevention of migraine: The multicenter, randomized, double-blind, sham-controlled PREMIUM II trial. Cephalalgia. 2022 Jun;42(7):560-569. doi: 10.1177/03331024211068813. Epub 2022 Jan 9. PMID 35001643